CLINICAL TRIAL: NCT01791062
Title: Safety and Efficacy of a Novel, Cell-free Cartilage Repair Construct in the Treatment of Focal Chondral Defects Involving the Femoro-tibial Compartment of the Knee Joint.
Brief Title: Safety and Efficacy Study of HYTOP® in the Treatment of Focal Chondral Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAREKT-DE-2011-12
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Focal Chondral Defect in Femoro-tibial Compartment of the Knee Joint
Keywords: cartilage tissue engineering; hyaluronan; hyaluronic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HYTOP® (Experimental)
  Interventions: Device: HYTOP®

INTERVENTIONS:
Device: HYTOP® — HYTOP® will be implanted once during surgery.

SUMMARY:
The two-layer bioresorbable HYTOP® matrix consists of an upper layer of highly purified porcine splint-skin which contains natural pores, and a lower layer of highly purified collagen fleece containing hyaluronan (HA).

In this study, the medical device will be used and evaluated in a one-step procedure combining microfracturing with surgical implantation of HYTOP®. HYTOP® will support haemostasis in the articular cartilage defect, act as a support for cell growth and as a three-dimensional scaffold for cell differentiation. HYTOP® will protect the underlying tissue after cartilage debridement and/or microfracturing of the subchondral bone.

The primary working hypothesis is that HYTOP® is safe and suitable as a cell-free matrix to support haemostasis, as a cover for the cartilage lesion and eventually to enhance cartilage regeneration in a one-step surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 50 years of age.
* Good general health condition.
* Signed written informed consent.
* General anaesthesia is justifiable for the patient from the medical point of view.
* Focal chondral defects involving the femorotibial compartment of the knee joint localised in only one compartment and not larger than the size of one HYTOP® patch.
* Isolated one-sided chondral lesion.
* Cartilage defect classified as Outerbridge grade 3 or 4.
* Chondral lesions not exceeding through the subchondral bone (intact subchondral bone).
* Nearly intact chondral structure surrounding the defect, specifically Outerbridge grade 2 or less.
* Corresponding joint area classified with maximum Outerbridge grade 2.
* Clinical symptoms in the target joint (pain on walking 100 m of more than 4 on an 11-point numerical scale or swelling or locking or 'giving way').
* Ensured compliance of subjects over the whole study period.

Exclusion Criteria:

* Treatment with any investigational product within 4 weeks prior to study entry.
* Patients with known hypersensitivity to the constituents of the product or any component or procedure used in the study.
* Patients with previous treatment of the study relevant defect site.
* Cartilage lesion is not intact shouldered, has bipolar or corresponding involvement or bipolar 'kissing' lesions.
* Necessity of cartilage repair treatment at bilateral joints.
* Patients with meniscus lesions, total or partial (more than 1/3 of total volume) resected meniscus, limited joint mobility, varus/valgus joint malalignment of more than 5 degrees or insufficient ligament support.
* Inflammatory joint diseases (e.g. rheumatoid arthritis, Bechterew disease, chondromatosis).
* Infection at study relevant site.
* Osteoarthritis, arthrofibrosis or haematopoetic related diseases.
* Study relevant metabolic disease, adipositas (BMI equal to or greater 30 kilogram per square meter).
* Study relevant neoplastic, neurological or mental illness.
* Study relevant autoimmune disease.
* Patients with elevated risk of bleeding.
* Recent history of drug and/or alcohol abuse (within the last 6 months).
* Pregnant or lactating females.
* Participants of childbearing age (pre-menopausal) who do not accept the use of methods of birth control with pearl index more than 1% (e.g. oral contraceptives, vaginal ring, hormone-releasing intrauterine device (IUD), implants, depot syringes, hormone patch, double barrier method, tubal ligation, vasectomised partner,…) during the treatment period and the first 12 weeks of follow-up period.
* Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and/or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language).
* Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts.
* Low probability of compliance with after-care rehabilitation scheme.
* Forbidden concomitant treatment affecting the evaluation of study parameters (e.g. oral intake of chondroitin sulfate, glucosamine, piascledine, other i.a. treatments like depot corticosteroids or arthroscopic procedures).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events with causal relationship to the investigational medical device. | Up to 2 years (plus or minus 14 days) after surgery.
  Adverse events with causal relationship to the investigational medical device (judged as 'related', 'possibly related' or 'relationship not assessable') will be evaluated with respect to type, incidence and intensity up to study termination of each subject.

SECONDARY OUTCOMES:
All adverse events without causal relationship to the investigational medical device. | Up to 2 years (plus or minus 14 days) after surgery.
  Adverse events without causal relationship to the investigational medical device (judged as 'not related') will be evaluated with respect to type, incidence and intensity up to study termination of each subject.
Joint girth measurement | Baseline
  Knee girth measurement as a marker for swelling is taken around the knee at the level of mid-patella as well as 10 centimeters (cm) proximal and distal and documented in cm.
Joint girth measurement | On Day 180 (plus or minus 14 days) after surgery.
  Knee girth measurement as a marker for swelling is taken around the knee at the level of mid-patella as well as 10 centimeters (cm) proximal and distal and documented in cm.
Joint girth measurement | On Day 360 (plus or minus 14 days) after surgery.
  Knee girth measurement as a marker for swelling is taken around the knee at the level of mid-patella as well as 10 centimeters (cm) proximal and distal and documented in cm.
Joint girth measurement | On Day 5 after surgery.
  Knee girth measurement as a marker for swelling is taken around the knee at the level of mid-patella as well as 10 centimeters (cm) proximal and distal and documented in cm.
Pain intensity | Baseline
  Intensity of pain on walking 100 meters will be evaluated on 11-point ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Pain intensity | On Day 180 (plus or minus 14 days) after surgery.
  Intensity of pain on walking 100 meters will be evaluated on 11-point ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Pain intensity | On Day 360 (plus or minus 14 days) after surgery.
  Intensity of pain on walking 100 meters will be evaluated on 11-point ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Pain intensity | On Day 5 after surgery.
  Intensity of pain on walking 100 meters will be evaluated on 11-point ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
Magnetic Resonance Imaging (MRI) Signal intensity | On Day 180 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to signal intensity of the cartilage repair tissue as 'not isointense', 'isointense' or 'not assessable'.
MRI Signal intensity | On Day 360 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to signal intensity of the cartilage repair tissue as 'not isointense', 'isointense' or 'not assessable'.
Presence of lesions | On Day 180 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to lesions in the cartilage repair tissue as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of lesions | On Day 360 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to lesions in the cartilage repair tissue as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone oedema | Baseline
  MRI will be assessed with respect to presence of subchondral bone oedema as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone oedema | On Day 180 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone oedema as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone oedema | On Day 360 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone oedema as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone cyst | Baseline
  MRI will be assessed with respect to presence of subchondral bone cyst as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone cyst | On Day 180 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone cyst as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone cyst | On Day 360 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone cyst as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of effusion | Baseline
  MRI will be assessed with respect to presence of effusion as 'no', 'yes' or 'not assessable'.
Presence of effusion | On Day 180 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of effusion as 'no', 'yes' or 'not assessable'.
Presence of effusion | On Day 360 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of effusion as 'no', 'yes' or 'not assessable'.
Joint girth measurement | On Day 720 (plus or minus 14 days) after surgery.
  Knee girth measurement as a marker for swelling is taken around the knee at the level of mid-patella as well as 10 centimeters (cm) proximal and distal and documented in cm.
Pain intensity | On Day 720 (plus or minus 14 days) after surgery.
  Intensity of pain on walking 100 meters will be evaluated on 11-point ordinal scale ranging from '0' (no pain) to '10' (extreme pain).
MRI Signal intensity | On Day 720 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to signal intensity of the cartilage repair tissue as 'not isointense', 'isointense' or 'not assessable'.
Presence of lesions | On Day 720 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to lesions in the cartilage repair tissue as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone oedema | On Day 720 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone oedema as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of subchondral bone cyst | On Day 720 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of subchondral bone cyst as 'absent', 'minimal', 'moderate', 'severe' or 'not assessable'.
Presence of effusion | On Day 720 (plus or minus 14 days) after surgery.
  MRI will be assessed with respect to presence of effusion as 'no', 'yes' or 'not assessable'.
Knee injury and osteoarthritis outcome score (KOOS) | Baseline
  The KOOS score consists of five separate scores calculated for pain, symptoms, activities of daily living, sport and recreational function and knee-related quality of life. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The results can be plotted as an outcome profile.
Knee injury and osteoarthritis outcome score (KOOS) | On Day 5 after surgery.
  The KOOS score consists of five separate scores calculated for pain, symptoms, activities of daily living, sport and recreational function and knee-related quality of life. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The results can be plotted as an outcome profile.
Knee injury and osteoarthritis outcome score (KOOS) | On Day 180 (plus or minus 14 days) after surgery.
  The KOOS score consists of five separate scores calculated for pain, symptoms, activities of daily living, sport and recreational function and knee-related quality of life. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The results can be plotted as an outcome profile.
Knee injury and osteoarthritis outcome score (KOOS) | On Day 360 (plus or minus 14 days) after surgery.
  The KOOS score consists of five separate scores calculated for pain, symptoms, activities of daily living, sport and recreational function and knee-related quality of life. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The results can be plotted as an outcome profile.
Knee injury and osteoarthritis outcome score (KOOS) | On Day 720 (plus or minus 14 days) after surgery.
  The KOOS score consists of five separate scores calculated for pain, symptoms, activities of daily living, sport and recreational function and knee-related quality of life. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The results can be plotted as an outcome profile.
Subjective knee evaluation form | Baseline
  The Subjective knee evaluation form of the International Knee Documentation Committee (IKDC) is used to assess symptoms, knee function and sporting activities in patients. The form consists of 18 questions in the domains of symptoms, functioning during activity of daily living and sports, current function of the knee, and participation in work and sports.
Subjective knee evaluation form | On Day 5 after surgery.
  The Subjective knee evaluation form of the International Knee Documentation Committee (IKDC) is used to assess symptoms, knee function and sporting activities in patients. The form consists of 18 questions in the domains of symptoms, functioning during activity of daily living and sports, current function of the knee, and participation in work and sports.
Subjective knee evaluation form | On Day 180 (plus or minus 14 days) after surgery.
  The Subjective knee evaluation form of the International Knee Documentation Committee (IKDC) is used to assess symptoms, knee function and sporting activities in patients. The form consists of 18 questions in the domains of symptoms, functioning during activity of daily living and sports, current function of the knee, and participation in work and sports.
Subjective knee evaluation form | On Day 360 (plus or minus 14 days) after surgery.
  The Subjective knee evaluation form of the International Knee Documentation Committee (IKDC) is used to assess symptoms, knee function and sporting activities in patients. The form consists of 18 questions in the domains of symptoms, functioning during activity of daily living and sports, current function of the knee, and participation in work and sports.
Subjective knee evaluation form | On Day 720 (plus or minus 14 days) after surgery.
  The Subjective knee evaluation form of the International Knee Documentation Committee (IKDC) is used to assess symptoms, knee function and sporting activities in patients. The form consists of 18 questions in the domains of symptoms, functioning during activity of daily living and sports, current function of the knee, and participation in work and sports.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Engelhardt, Dr., Principal Investigator — Klinikum Osnabrück GmbH Finkenhügel, Klinik für Orthopädie, Unfall- und Handchirurgie, Osnabrück (Germany)
Locations (1):
- Klinikum Osnabrück GmbH Finkenhügel, Klinik für Orthopädie, Unfall- und Handchirurgie, Osnabrück, Lower Saxony, Germany